CLINICAL TRIAL: NCT05788614
Title: In a Reverse Shoulder Arthroplasty, Does Function Depend on the Humeral Version? A Prospective Randomized Study.
Brief Title: Retroversion in Reverse Shoulder Arthroplasty
Acronym: RV-RSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, José Carlos Minarro, Principal investigator, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUReinaSofia
Record Dates: First submitted 2023-03-14; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RSA-RV-30 (Experimental)
  Interventions: Device: Reverse shoulder arthroplasty
- RSA-RV-0 (Experimental)
  Interventions: Device: Reverse shoulder arthroplasty

INTERVENTIONS:
Device: Reverse shoulder arthroplasty — Reverse shoulder arthroplasty

SUMMARY:
The goal of this clinical trial is to compare function in reverse shoulder arthroplasty (RSA) using two different degrees of humeral retroversion (RV). The main question it aims to answer is:

• Does external rotation improves when using a higher retroversion?

Participants will randomly receive a 0 degree or 30 degree RV for their RSA.

They will be followed for two years and clinical outcomes will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients > 60 years
* primary rotator cuff arthropathy
* implantation of reverse shoulder arthroplasty

Exclusion Criteria:

* previous surgeries in the shoulder
* post-traumatic arthropathy

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
External rotation of the shoulder | 2 years
  External rotation of the shoulder will be measured in degrees with the help of a goniometer in two ways.
  First: External rotation 1 (ER1): arm adducted at zero degrees Second: External rotation 2 (ER2): arm in 90 degrees of abduction.
Constant-Murley Score | 2 years
  The Constant-Murley score is a multi-item functional scale assessing pain, daily activities, range of motion and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos Minarro, Dr, Principal Investigator — Hospital Universitario Reina Sofía de Córdoba
Locations (1):
- Hospital Universitario Reina Sofía de Córdoba, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided